CLINICAL TRIAL: NCT02010788
Title: Evaluation of Safety and Efficacy of Botulinum Toxin Type A (BOTOX®) to Treat Urinary Incontinence Due to Neurogenic Detrusor Overactivity or Overactive Bladder in Korea
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 191622-134
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Urinary Incontinence; Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BOTOX®: Patients who receive botulinum toxin Type A (BOTOX®) treatment for Neurogenic Detrusor Overactivity or Overactive Bladder as per local standard of care in clinical practice.
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — Botulinum toxin Type A treatment for Neurogenic Detrusor Overactivity or Overactive Bladder as per local standard of care in clinical practice.
  Other Names: BOTOX®; onabotulinumtoxinA

SUMMARY:
This study is a Post-Marketing Surveillance study in Korea to evaluate the safety and efficacy of botulinum toxin Type A to treat urinary incontinence in patients with neurogenic detrusor overactivity (NDO) or overactive bladder (OAB) not adequately controlled by anticholinergic drugs.

ELIGIBILITY:
Inclusion Criteria:

-Patients with urinary incontinence due to NDO or OAB treated with BOTOX® as per local standard of care in clinical practice.

Exclusion Criteria:

-None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with urinary incontinence due to NDO or OAB.
Sampling Method: Non-Probability Sample
Enrollment: 523 (Actual)
Dates: Start 2014-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events and Adverse Drug Reactions | 4 Months
International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) Total Score | 4 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com